CLINICAL TRIAL: NCT04253548
Title: Implementation and Effectiveness Evaluation of the iPeer2Peer Support Mentorship Program Within Pediatric Thoracic Transplantation
Brief Title: iPeer2Peer Pediatric Thoracic Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Enduring Hearts (Unknown); University of Alberta/Stollery Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Samantha Anthony, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000065141
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Solid Organ Transplant
Keywords: Peer Support Mentorship; Transplant; Pediatrics; Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPeer2Peer Program (Experimental): Participates in the iPeer2Peer Program
  Interventions: Behavioral: iPeer2Peer Support Mentorship Program

INTERVENTIONS:
Behavioral: iPeer2Peer Support Mentorship Program — iPeer2Peer is an online peer support mentorship program that has been established in multiple chronic disease populations as a self-management intervention, including chronic pain and juvenile idiopathic arthritis. The iPeer2Peer program provides modeling and reinforcement by pre-screened and trained young adult peer mentors to adolescent mentees.

SUMMARY:
With the on-going presence of a chronic illness, daily immunosuppressive medications, and the need for continuous medical supervision, pediatric transplant recipients face considerable psychosocial stresses. Treatment nonadherence is a major issue in pediatric transplantation and can lead to increased rates of hospitalization, rejection episodes, graft loss and death. An online peer support mentorship program (iPeer2Peer) is proposed as one intervention that could enhance patient care management, increase treatment adherence, reduce social isolation and improve health outcomes for this highly vulnerable population. The proposed trial will determine 1) implementation outcomes of the iPeer2Peer intervention in terms of: (a) feasibility and adoption, (b) acceptability and appropriateness and (c) level of engagement with the program, and 2) effectiveness of the iPeer2Peer intervention on improving health outcomes including disease self-management skills, treatment adherence, quality of life, perceived social support, stress and coping.

ELIGIBILITY:
Inclusion Criteria:

1. heart and/or lung transplant recipient,
2. at least 4 months post-transplant,
3. between the ages of 12 and 25 years,
4. able to speak and read English,
5. willingness to commit to 5-10 texts and/or calls of 20-30 minutes each over a period of 15 weeks.

Exclusion Criteria:

1. have a significant cognitive impairments as assessed by a qualified healthcare provider,
2. have a diagnosis of an active psychological disorder (e.g., Major Depressive Disorder, Generalized Anxiety Disorder) likely to influence assessment of health-related quality of life and/or interfere with their ability to manage their transplant regimen (a diagnosis of an active psychological disorder will be determined for mentees through medical chart review and self-reported by mentors), and
3. are participating in other peer support or self-management interventions

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability: Semi-structured Interview (Mentees) | 15 weeks after baseline/immediately after the intervention
  Semi-structured Interview
Acceptability: Semi-structured Interview (Mentors) | Study completion, an average of 1 year
  Semi-structured Interview
Adoption (Mentees) | 15 weeks after baseline/immediately after the intervention
  Semi-structured Interview
Adoption (Mentors) | Study completion, an average of 1 year
  Semi-structured Interview
Adoption | Mentees - 12 weeks post-program completion; Mentors - study completion, an average of 1 year
  Accrual and dropout rates
Adoption | Mentees - 12 weeks post-program completion; Mentors - study completion, an average of 1 year
  Compliance with iPeer2Peer program
Feasibility: Semi-structured Interview (Mentees) | 15 weeks after baseline/immediately after the intervention
  Semi-structured Interview
Feasibility: Semi-structured Interview (Mentors) | Study completion, an average of 1 year
  Semi-structured Interview
Feasibility: Accrual and dropout rates | Mentees - 12 weeks post-program completion; Mentors - study completion, an average of 1 year
  Accrual and dropout rates
Feasibility: Compliance with iPeer2Peer program (Mentees) | 12 weeks post-program completion
  Compliance with iPeer2Peer program (an 80% rate of completion of five calls and online outcome measures)
Feasibility: Compliance with iPeer2Peer program (Mentors) | Study completion, an average of 1 year
  Compliance with iPeer2Peer program (an 80% rate of completion of five calls and online outcome measures)
Appropriateness (Mentees) | 15 weeks after baseline/immediately after the intervention
  Semi-structured Interview
Appropriateness (Mentors) | Study completion, an average of 1 year
  Semi-structured Interview
Level of Engagement (Mentees) | 15 weeks after baseline/immediately after the intervention
  Semi-structured Interview
Level of Engagement (Mentors) | Study completion, an average of 1 year
  Semi-structured Interview

SECONDARY OUTCOMES:
Disease self-management skills (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Self-management skills assessment guide (questionnaire); 21-item questionnaire. Each question is scored on a scale from 1 to 5.
Treatment adherence (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Adolescent Medication Barriers Scale; 17-item questionnaire with 3 different sections: Disease Frustration/Adolescent Issues, Ingestion Issues, and Regimen Adaptation/Cognitive. Each question is scored on a scale from 1 to 5. An overall higher score means a worse outcome.
Treatment adherence (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Immunosuppressant Blood Levels
Treatment adherence (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Clinic Attendance
Quality of Life (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Pediatric Quality of Life Inventory™ 3.0 Transplant Module; 46-item questionnaire with 8 different sections: About My Medicines I, About My Medicines II, My Transplant and Others, Pain and Hurt, Worry, Treatment Anxiety, How I Look, and Communication. Each question is scored on a scale from 0 to 4. An overall higher score means a better outcome.
Perceived Social Support (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  National Institute of Health Emotional Support Survey; 7-item questionnaire. Each question is scored on a scale from 1 to 5. An overall higher score means a better outcome.
Emotional Distress (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Revised Child Anxiety and Depression Scale - short version; 25-item questionnaire. Each question is scored on a scale with 4 possible responses. An overall higher score means a worse outcome.
Resiliency (Mentees) | Baseline, 15 weeks after baseline/immediately after the intervention, 12 weeks post-program completion
  Brief Resilience Scale; 6-item questionnaire. Each question is scored on a scale with 5 possible responses. An overall higher score means a better outcome.
Quality of Mentor Behaviour (Mentees) | 15 weeks after baseline/immediately after the intervention
  Mentor Behaviour Scale; 15-item questionnaire with 4 different sections: Structure, Engagement, Autonomy Support, and Competency Support. Each question is scored on a scale from 1 to 5.
Change in Physical and Emotional Symptoms (Mentors) | Baseline, pre-intervention; study completion, an average of 1 year
  PROMIS - 29 Adult Profile v2.1; Maximum 29-item questionnaire as responses to some questions may lead participants to answer fewer questions. There are 8 different sections: Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity. Each question is scored on a scale from 1 to 5.
Change in Perceived Social Role Satisfaction (Mentors) | Baseline, pre-intervention; study completion, an average of 1 year
  PROMIS Satisfaction with Social Roles and Activities; Maximum 44-item questionnaire as responses to some questions may lead participants to answer fewer questions. Each question is scored on a scale from 1 to 5. An overall higher score means a better outcome.
Change in Self-efficacy (Mentors): Chronic Disease Self-Efficacy Scale | Baseline, pre-intervention; study completion, an average of 1 year
  Chronic Disease Self-Efficacy Scale; 33-item questionnaire with 10 different sections: Exercise Regularly Scale, Get Information About Disease Item, Obtain Help from Community/Family/Friends Scale, Communicate With Physician Scale, Manage Disease in General Scale, Do Chores Scale, Social/Recreational Activities Scale, Manage Symptoms Scale, Manage Shortness of Breath Item, and Control/Manage Depression Scale. Each question is scored on a scale from 1 to 10. An overall higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Anthony, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No